CLINICAL TRIAL: NCT02450162
Title: Comparison of the Changes of Lateral Rectus Muscle Insertion Measured With AS-OCT in Two Recession Surgeries
Brief Title: Lateral Rectus Muscle and Anterior Segment Optical Coherence Tomography (AS-OCT) in Two Recession Surgeries
Acronym: AS-OCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-02-115
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-04

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- conventional lateral rectus recession: This is the standard technique for recession with two single-armed sutures.Exposure of the rectus muscle insertion includes freeing the insertion and proximal muscle borders sufficiently to place the sutures. And the needle is passed through the tendon avoiding the anterior ciliary arteries. If the sutures are passed as shown a true knot is formed, and the muscle is detached. Then a caliper measures from the limbus or the original insertion. A passage of the needle through sclera. The recessed muscle is ideally parallel to the old insertion (or nearly so). Conjunctival incision was finally sutured.
  Interventions: Procedure: lateral rectus recession (bilateral)
- hang-back lateral rectus recession: The hang-back recession has been described as "a simple, safe alternative to conventional recession." The procedure is said to be less likely to result in scleral perforation because needles are placed through relatively thicker sclera near the insertion site. It is the modified techique for recession with one double-armed sutures.
  Interventions: Procedure: lateral rectus recession (bilateral)

INTERVENTIONS:
Procedure: lateral rectus recession (bilateral) — Two types of recession (conventional or hang-back method) are typical surgeries for correcting intermittent exotropia. It depends on surgeon's decision at the time of surgery.

SUMMARY:
* Background and study aims : The investigators conducted this study to compare the movement of extraocular muscle after two types of recession surgery with non-invasive tool called AS-OCT.
* Who can participate? patients who will undergo two types (conventional method and hang-back method) of typical bilateral lateral rectus recession surgery for correcting intermittent exotropia
* What does the study involve? Volunteers will attend a clinic for four visits over three months. They will undergo AS-OCT at every visits during follow up period. AS-OCT is non-invasive test to evaluate operation site. The test only requires their cooperation when they undergo AS-OCT.
* What are the possible benefits and risks of participating? This is non-invasive test for your postoperative follow up. Therefore, there will be no risks about this test.
* Where is the study run from? Samsung Medical Center
* When is the study starting and how long is it expected to run for? From April 2015 to Dec 2015

DETAILED DESCRIPTION:
This study is a following study of our prior study about AS-OCT in strabismus. The aim of this study is to compare the longitudinal changes of lateral rectus (LR) muscle insertion between two types of bilateral recession surgery. An AS-OCT scan of the LR muscle was performed every visits. Data on gender, age, degree of deviation (prism diopter), and spur-LR insertion distance using AS-OCT were collected at postoperative months 1,3 in each group.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo bilateral lateral rectus recession surgery for correcting intermittent exotropia

Exclusion Criteria:

* previous ocular surgery
* other ocular diseases except intermittent exotropia
* amblyopia

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 60 patients
  : 30 for conventional recession surgery 30 for hang-back recession surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The change of limbus-muscle insertion distance measured with AS-OCT | baseline and 1.3 months